CLINICAL TRIAL: NCT04018898
Title: Older Emergency Department Users and Short-term Adverse Events at the Index Visit: Which Clinical Prognostic Tool is Used?
Brief Title: Older Emergency Department Users and Short-term Adverse Events at the Index Visit
Status: Completed | Type: Observational
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Olivier Beauchet, MD, Professor of Geriatrics, Jewish General Hospital
Other Study IDs: 2020-1881
Record Dates: First submitted 2019-07-11; First posted 2019-07-15 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Health Impairment; Adverse Event; Hospitalization

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: Each participant will be evaluated at Emergency Department based on ER2 screening tool (Emergency Room Evaluation and Recommendation Form). Six closed-ended format questions (i.e., yes versus no) composed ER2 assessment: Age category (≥ 85), male, polypharmacy (≥ 5 different medications per day), use of formal (health care or social professional) and/or informal (family and/or friend) home support, use of a walking aid regardless its type, and temporal disorientation (inability to give the current month and/or year).

SUMMARY:
This study evaluates the difference between PRISMA-7 and ER2 tool. There are some differences between PRISMA-7 and ER2 tool. The differences consist in evaluation criteria that are used to perform the both surveys. We suppose that evaluation criteria of PRISMA-7 is not accurately enough to calculate the length of hospital stay and to predict the short-term outcomes.

DETAILED DESCRIPTION:
The "Program of Research on Integration of Services for the Maintenance of Autonomy" (PRISMA-7) is the Ministry of Health and Social Services' reference tool for the assessment of older ED users in Quebec (Canada). PRISMA-7 has been initially designed to screen disability in community-dwelling older adults and has never been validated for risk for short-term adverse events in older ED users. "Emergency room evaluation and recommendations" (ER2) is another clinical tool which is currently evaluated in Quebec. Compared to PRISMA-7, ER2 has been especially designed for assessing risk for short-term ED adverse events. No study has compared PRISMA-7 and ER2 risk for short-term adverse events. We hypothesised that ER2 could be a better prognostic tool compared to PRISMA-7 for long length of stay in ED and hospital stay, and hospital admission because it was designed and validated for this specific goal. The study aims to 1) examine and compared PRISMA-7 and ER2 risk for long length of ED and hospital stay and hospital admission, and 2) to establish their performance criteria (i.e., sensitivity, specificity, positive predictive value, negative predictive value, likelihood ratios) for these three short-term adverse events in older ED users.

ELIGIBILITY:
Inclusion Criteria:

* Being 75 years old and over
* Brought at Emergency on medical stretcher

Exclusion Criteria:

* Being less than 75 years old
* Never come at Emergency

Min Age: 75 Years | Sex: All
Age Groups: Older Adult
Study Population: In this study will be enrolled people who are 75 years and over, and who come at Emergency not only for medical reason but also for social.
Sampling Method: Non-Probability Sample
Enrollment: 10971 (Actual)
Dates: Start 2019-07-23 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Short-term adverse events | Around 10 months
  The adverse event is defined as an adverse outcome related to an ED encounter, this adverse event is related to ED care.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Beauchet, MD, Principal Investigator — Jewish General Hospital
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada